CLINICAL TRIAL: NCT00471367
Title: A Phase I, Open-Label, Multi-Center, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD4877 Administered Twice a Week in Adult Patients With Advanced Solid Malignancies Including Lymphoma
Brief Title: Phase I, Open-label, Dose-escalation, Safety and PK Study of AZD4877
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part B of the study was terminated early due to a lack of enrollment.
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2782C00006
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2009-09

CONDITIONS: Lymphoma; NHL; Non-Hodgkin Lymphoma
Keywords: Phase I; AZD4877; Lymphoma; B-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — N-(3-aminopropyl)-N-(1-(5-benzyl-3-methyl-4-oxo-(1,2)thiazolo(5,4-d)pyrimidin-6-yl)-2-methylpropyl)-4-methylbenzamide

INTERVENTIONS:
Drug: AZD4877 — intravenous infusion administered twice a week for 2 weeks

SUMMARY:
This study has two parts (A and B). The primary purpose of Part A is to find the maximum tolerated dose is for an experimental drug called AZD4877 based on the side effects experienced by patients that receive AZD4877 on a twice a week basis. For Part B, an additional 20 patients will be treated at the maximum dose identified in Part A. AZD4877 is an Eg5 or Kinesin Spindle Protein inhibitor that interferes with tumor cell division leading to tumor growth

ELIGIBILITY:
Inclusion Criteria:

* Part A: Advanced solid tumors (including lymphoma without bone marrow involvement) for which standard treatment doesn't exist or is no longer effective.
* Part B: B-cell non-Hodgkin lymphoma that is not eligible for curative therapy or has relapsed.
* Relatively good overall health other than your cancer

Exclusion Criteria:

* Poor bone marrow function (not producing enough blood cells). Serious heart conditions. Poor liver or kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-04; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To identify a maximum tolerated dose of AZD4877 by assessment of the incidence of dose limiting toxicities | on a twice a week schedule for two weeks out of every three weeks

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of AZD4877 by assessment of Common Terminology Criteria for Adverse Events version 3.0 (CTCAE) grade and type of AE, changes in laboratory values, vital signs, and incidence of protocol defined dose modification | assessed after each course of treatment
Dose Expansion (Part B):Estimate efficacy of AZD4877 through evaluation of objective response rate, progression-free survival and disease control rate in patients with B-cell non-Hodgkin lymphoma using the revised response criteria for malignant lymphoma | Assessed during treatment and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — AstraZeneca; Lea Burke, Study Chair — AstraZeneca
Locations (3):
- United States (3):
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina